CLINICAL TRIAL: NCT00729560
Title: Determination if Pharmacologic Blockade of Androgen Action Decreases Renal Clearance of D-Chiro-Inositol (DCI), Increases the Circulating Concentration of DCI, and Enhances Insulin-Stimulated Release of the D-chiro-inositol-containing Inositolphosphoglycan (DCI-IPG) Mediator in Obese Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Effects of Flutamide on Insulin and Glucose Metabolism in Women With Polycystic Ovary Syndrome
Acronym: PCOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 04487VCUIRB; GCRC0826
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Flutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Flutamide
  Interventions: Drug: Flutamide
- 2 (Placebo Comparator): control to arm 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flutamide — 250 mg twice daily for 4 weeks
  Arms: 1
Drug: Placebo — Placebo twice daily for 4 weeks
  Arms: 2

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is the major cause of infertility in the United States. Many women with PCOS demonstrate insulin resistance and a compensatory hyperinsulinemia.This is due to both an intrinsic form of insulin resistance unique to PCOS and, in many cases, acquired insulin resistance due to obesity. The importance of this observation lies in the fact that hyperinsulinemia appears to play an important pathogenetic role in the hyperandrogenism and anovulation of both obese and lean women with PCOS.

DETAILED DESCRIPTION:
Hyperinsulinemia stimulates ovarian production of androgens, especially testosterone, in PCOS. Therefore, it is theoretically possible that testosterone increases urinary clearance of D-chiro-inositol (uCl(DCI) in PCOS, and that this serves as the explanation for the correlation between uClDCI and insulin sensitivity. While we regard this possibility as unlikely, it is important that it be tested. To accomplish this, we will assess obese (Body Mass Index (BMI) >30 kg/m2) women with and without PCOS at baseline, and again after 4 weeks of androgen action blockade with the drug flutamide. Flutamide is an antiandrogen that works by blocking the binding of androgens to the androgen receptor.

We will determine if this pharmacologic blockade i) decreases the renal clearance of DCI, ii) increases the circulating concentration of DCi, and iii) enhances the insulin-stimulated release of the D-chiro-inositol-containing inositolphosphoglycan (DCI-IPG) mediator during an OGTT.

ELIGIBILITY:
Inclusion Criteria:

(1) Obese (BMI≥30 kg/m2) women with PCOS between 18-40 years of age: i) oligomenorrhea (8 menstrual periods annually), ii) biochemical hyperandrogenemia (elevated total or free testosterone), iii) normal thyroid function tests and serum prolactin, and iv) exclusion of 21α-hydroxylase deficiency by a fasting 17α-hydroxyprogesterone <200 ng/dl.48, (2) acceptable health on the basis of interview, medical history, physical examination, and laboratory tests (complete blood chemistry (CBC), complete metabolic panel (CMP), urinalysis, serum Beta-Human Chorionic Gonadotropin (BhCG)). (3) Signed, witnessed informed consent. (4) Ability to comply with study requirements.

Exclusion Criteria:

(1) Diabetes mellitus by fasting glucose or oral glucose tolerance test (OGTT), or clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, neoplastic and malignant disease (other than non-melanoma skin cancer). (2) Current use of oral contraceptives. (3) Documented or suspected recent (within one year) history of drug abuse or alcoholism. (4) Ingestion of any investigational drug within two months prior to study onset.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Nestler, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University General Clinical Research Center, Richmond, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.vcu.edu/pcos

RESULTS

PARTICIPANT FLOW:
Groups:
- Flutamide and Placebo Control Subjects: Number of participants randomized to each Arm/Group is unknown, study was terminated before unblinding and no key exists.
Period: Overall Study
Arm/Group | Flutamide and Placebo Control Subjects
Started | 8 (Arm assignment can not be determined as study was ended prior to unblinding and no key found.)
Completed | 5
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Flutamide Treated and Placebo Control: Flutamide treated: 250 mg twice daily for 4 weeks or Placebo control: twice daily for 4 weeks. Study was terminated due to insufficient enrollment. Randomization is unknown as study was terminated prior to unblinding and no key can be found. Consequently, we are unable to differentiate between treated and control subjects.
Arm/Group | Flutamide Treated and Placebo Control
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: DCI-IPG Measurements in Blood and Urine
Description: zero participants analyzed, no assays performed
Time Frame: 2 years
Arm/Group | Flutamide and Placebo Control Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Flutamide Treated and Placebo Control Subjects: Flutamide: 250 mg twice daily for 4 weeks or Placebo: twice daily for 4 weeks
Arm/Group | Flutamide Treated and Placebo Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No